CLINICAL TRIAL: NCT00493389
Title: Improving The Assessment of Hypothalamic Pituitary Adrenal Function In Acute Stress
Brief Title: Cortisol Response to Adrenocorticotrophin (ACTH) in Acute Stress
Acronym: CRAAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Dr T C Ooi, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007255-01H
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-07

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: ACTH stimulation test; cortisol; stress
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Adrenocorticotrophic hormone

SUMMARY:
Cortisol deficiency is diagnosed by the adrenocorticotrophin (ACTH) stimulation test. This test measures cortisol levels in the blood before and after giving an injection of ACTH. Currently, the results of this test can only be reliably interpreted when it is carried out on people in non-stressful situations. Frequently the test is carried out in hospitalized patients in stressful situations, giving results that are hard to interpret.

Our study is to first do this test in a non-stressful situation, followed by a repeat test in a stressful situation, to compare the results and create a set of guidelines for interpreting the test when it is carried out in stressful situations.

DETAILED DESCRIPTION:
This study proposes to provide the reference range of cortisol results when the ACTH stimulation test is done under stressful conditions. This important information is currently not available in the literature. To achieve this, we will perform the ACTH stimulation test in a cohort of patients who are booked for elective surgery. By choosing elective surgery patients, we afford ourselves the opportunity of performing the test once before surgery. The test is then repeated within 12 hours of surgery. The first test will be done on an out-patient basis under usual conditions (minimal stress) while the second will be done under intense physical stress. The 2 sets of results will be compared and the effect of stress on test results will be determined. For the sake of uniformity, we have chosen patients who are booked to undergo repair of an abdominal aortic aneurysm (AAA) as our study cohort.

The ACTH stimulation is an important test that suffers from limitations resulting from lack of clear guidelines for the interpretation of results done under stressful conditions. This study will thus improve the usefulness of an important tool in the evaluation of the hypothalamic-pituitary-adrenal axis in stressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40 to 80 years, who are booked for elective open repair of abdominal aortic aneurysm at The Ottawa Hospital Civic campus

Exclusion Criteria:

* Inability to provide informed consent
* Pre-operative signs and symptoms of hypofunction of the HPA axis
* Pre-operative AST results that indicate HPA failure, necessitating perioperative hydrocortisone coverage (Cortisol level post-ACTH < 500 nmol/L)
* Presence of multiple co-morbidities such as poorly controlled diabetes, dialysis-dependant renal failure, hepatic failure
* Presence of hypoalbuminaemia < 35 g/L
* Untreated endocrine disorders such as hypothyroidism, hypopituitarism, hypogonadism detected by pre-operative measurement of TSH, FT4, LH, FSH and free testosterone. Such patients will receive any appropriate treatment prior to surgery. Once treated, participation in the study will be offered again and results analysed separately
* Being on drugs (a) that affect cortisol synthesis (eg. Ketoconazole, etomidate) or protein binding (eg. Estrogens), (b) any form of glucocorticoid which would inhibit CRH and ACTH secretion.
* Use of herbal or anabolic supplements

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
cortisol response | within 12 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Teik-Chye Ooi, MBBS, FRCPC,, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Riverside campus, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Streeten DH, Anderson GH Jr, Bonaventura MM. The potential for serious consequences from misinterpreting normal responses to the rapid adrenocorticotropin test. J Clin Endocrinol Metab. 1996 Jan;81(1):285-90. doi: 10.1210/jcem.81.1.8550765.
- [Background] Sibbald WJ, Short A, Cohen MP, Wilson RF. Variations in adrenocortical responsiveness during severe bacterial infections. Unrecognized adrenocortical insufficiency in severe bacterial infections. Ann Surg. 1977 Jul;186(1):29-33. doi: 10.1097/00000658-197707000-00005. PMID 195542
- [Background] Rothwell PM, Udwadia ZF, Lawler PG. Cortisol response to corticotropin and survival in septic shock. Lancet. 1991 Mar 9;337(8741):582-3. doi: 10.1016/0140-6736(91)91641-7. PMID 1671944
- [Derived] Druce I, Abujrad H, Chaker S, Meggison H, Hill A, Raymond A, Mayne J, Ooi TC. Circulating PCSK9 is lowered acutely following surgery. J Clin Lab Anal. 2018 May;32(4):e22358. doi: 10.1002/jcla.22358. Epub 2017 Nov 17. PMID 29148099